CLINICAL TRIAL: NCT03803592
Title: Effects of a Home Based, Dyadic Multisensory and Cognitive Stimulation (MCS) Program for the People With Dementia and Their Family Caregivers: a Pilot Quasi-experimental Study
Brief Title: Effect of a Dyadic Multisensory and Cognitive Stimulation Program for People With Dementia and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hong Kong Young Women's Christian Association (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Clinical Instructor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20180911003
Record Dates: First submitted 2018-10-19; First posted 2019-01-14 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Dementia; Carer Stress Syndrome
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: A two-arm non-randomized study design will be adopted to test the effect of a dyadic multisensory and cognitive stimulation program (MCS) for PWD and their caregivers between the intervention and control group. The Intervention group will attend the home-based dyadic MCS group, while the control group will receive the usual care. The dyadic MCS program is a 15-week program which composes of center-based face to face sessions (FTF) and caregiver-delivered home-based sessions. In the first 4 weeks, participants will attend the center-based FTF session twice a week (8 sessions), while in the remaining week (5th-15th Week), home-based sessions will be delivered by the caregivers at home and was suggested to deliver 3 times/week. To address any difficulties from the caregivers, the home-based sessions will be supplemented with weekly telephone follow-up and 2 FTF sharing sessions which will be held on the 8th and 12th week over the intervention period.
Who Masked: Outcomes Assessor
Masking Description: All outcome measurements will be collected by assessors who are blinded to the group assignment of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic MCS program (Experimental): Participants from the experimental group will receive a dyadic multisensory and cognitive stimulation (MCS) programme.
  The MCS program is a 15- week program. In the first 4 weeks, participants will attend the center-based Face-to-face (FTF) session twice a week (8 sessions), while in the remaining week (5th-15th Week), home-based sessions will be delivered by the caregivers with the PWD at home and was suggested to deliver the intervention 3 times/week at home. The home-based sessions will be supplemented with weekly telephone follow-up and two FTF sharing sessions over the intervention period.
  Interventions: Behavioral: Dyadic MCS program
- Control group (No Intervention): Participants from the control group will receive usual care and no intervention will be received.

INTERVENTIONS:
Behavioral: Dyadic MCS program — In the first 4 weeks, the dyads will attend the center-based FTF sessions. Each session will last for 1.5 hours. In the first 60 minutes, MCS activities (e.g. reality orientation, calculation and drawing) will be led by an occupational therapist. Skills in delivering the MCS activities will also be taught to equip CG with skills in leading the home-based sessions later. CG will leave in the last 30 minutes to attend a psychoeducation group on caregiving (led by social workers) and the PWD will continue the session.
  From week 5 onwards, The home based session (Week 5-15) will be delivered by the CG 3 times weekly at home (30 - 45min/ session).The sessions will be supplemented with weekly telephone follow-up and two FTF sharing sessions held on the 8th and 12th week over the period.
  Arms: Dyadic MCS program

SUMMARY:
Although multisensory and cognitive stimulation therapy was shown as an effective intervention in improving cognition and behavioral symptoms of people with dementia (PWD), it is not commonly found as an element in the previous dyadic interventions. It was believed that the involvement of the family caregivers in multisensory and cognitive stimulation therapy could produce additional benefits to both PWD and caregivers by enhancing their interactions. Therefore, we will conduct a pilot study which aims to explore the feasibility and the effects of a home based dyadic multisensory and cognitive stimulation (MCS) program for the PWD and their family caregivers followed by a randomized controlled trial (RCT). In the RCT, the intervention group will attend the home-based dyadic MCS group, while the control group will receive the usual care. The outcomes measurements of caregivers (positive caregiving experience, perceived stress, caregiver burden, and quality of life) and PWD (cognitive function and behavioral symptoms) will be assessed at baseline, immediately post intervention, and 3 month-follow up. To understand the therapeutic components and identify the strengths, limitations and difficulties of the home based dyadic MCS program, process evaluation will be conducted through semi-structured focus group interviews with 15 participants from the MCS group. It is hypothesized that the MCS group will have a significant improvement on positive caregiving experience, perceived stress, caregiver burden, and quality of life of caregivers and cognitive function and behavioral symptoms of PWD.

DETAILED DESCRIPTION:
Background:

Dementia becomes a major issue of worldwide concern. According to the World Alzheimer Report, the number of patients with dementia (PWD) worldwide was estimated at 46.8 million and it will be triply projected to 131.5 million in 2050. Similarly, dementia is also a prominent problem in Hong Kong. One in every three local seniors who are over 895 years of age suffered from dementia. The prevalence of PWD in Hong Kong will have a triple increase from 100,000 cases in 2009 to 300,000 cases in 2039.As the disease progresses, PWD will gradually lose their self-care ability and their cognitive function. In addition, behavioral symptoms such as agitation, delusion, and anxiety will appear on the sufferers. The caring burden and the uncertainty about the disease progress result in high levels of caring stress and negative emotion on family caregivers.

Nowadays, different psychosocial interventions have been designed for the PWD and their family caregivers to promote their psychological well-being. The dyadic intervention is deemed as one of the effective approach due to its mutual influence between the PWD and their family caregivers. A systematic review with 40 clinical trials found that dyadic approach can be integrated into different interventions such as psycho-education, and caring skills training . Although cognitive stimulation and multisensory stimulation therapy are regarded as an effective intervention for the cognition and the behavioral symptoms of the PWD, it is not commonly found as an element in the previous dyadic interventions. Involving family caregivers in a cognitive training can have some potential benefits for both caregivers and the PWD (e.g. cognitive function of the PWD and the quality of life) . The involvement of the family caregivers in the cognitive and multisensory stimulation therapy could promote the interactions between the PWD and caregivers which may produce additional benefits for both caregivers and the PWD, compared with the traditional cognitive stimulation therapy.

Objective:

The study aims to investigate the effects of the home based dyadic Multisensory and cognitive stimulation (MCS) intervention for the family caregivers of PWD in improving their positive aspects of caregiving, stress, depression, quality of life, and burden; and the cognitive function and behavioral symptoms of the PWD immediate post-intervention (T1) and, 3-month follow-up (T2), compared with the control group.

Methods:

A two- arm randomized controlled trial will be adopted to achieve the research objectives. After considering the number of group size and previous studies about the sample size, a total of 60 subjects (120 pairs of dyads-PWD and caregivers) will be recruited from four elderly community centers in Hong Kong with convenience sampling.

Participants from the Intervention group will attend the home-based dyadic MCS group, while the control group will receive the usual care. The outcomes measurements of caregivers (positive caregiving experience, perceived stress, caregiver burden, and quality of life) and PWD (cognitive function and behavioral symptoms) will be assessed by a blinded assessor at baseline (T0), immediately post intervention (T1) , and 3 month-follow up (T2). To understand the therapeutic components and identify the strengths, limitations and difficulties of the home based dyadic MCS program, process evaluation will be conducted through focus group interviews with 15 MCS participants after the intervention. In order to obtain a broad spectrum of views about the intervention, participants will be purposely selected for interview based on their level of stress reduction after the intervention.

IBM SPSS 23.0 will be used for the data analyses. Mixed multi-variate modeling or MANOVA test will be performed to investigate the between-group effect, the within-group effect (Times: T0, T1, and T2) and the interaction effect (Group x Time) on all of the outcomes variables. The last observation carried forward method will be adopted to replace the missing data if the missing value is in a small amount (<20%) and randomly distributed (Gray, Grove, & Burns, 2013; Hamer & Simpson, 2009). For the qualitative data, content analysis approach will be used to analyze all the transcribed interview verbatim.

Significance and Value:

The clinical project addresses the limitations of the previous psychosocial interventions and provides the PWD and their caregivers with an opportunity to improve the cognitive function of the PWD and promote the positive caregiving experience in the family caregivers which can reduce the caregivers' level of stress and improve the quality of life of the both family caregivers and the PWD. The findings from this projects can also inform the future direction in supporting the PWD and their family members and strengthen the nursing role in the community care.

ELIGIBILITY:
People with dementia and their family caregiver will be recruited.

The People with Dementia (PWD)

Inclusion Criteria:

* Aged 65 or above who had been diagnosed with any type of dementia,
* Community-dwelling (i.e., non-institutionalized)
* Understand Cantonese and able to follow simple instructions

Family Caregivers

Inclusion Criteria:

* Aged 18 years or above;
* The blood or by-marriage relatives (e.g. spouses, siblings, children, and grandchildren) of a person who has been clinically diagnosed with dementia, regardless of its types and these relatives are taking up the caring responsibilities ranging from physical aids to emotional supports, in the form of transportation, financial assistance, personal hygiene, and decision-making.;
* Providing most of the daily care and support for PWD (daily contact for at least four hours); and
* Able to speak Cantonese

Exclusion Criteria for PWD and their family caregivers:

* Diagnosed with a mental disorder such as bipolar disorder, schizophrenia, or depression; and/or,
* Currently taking anticonvulsants, or any kind of psychotropic drugs, and/or identified with a self-reported suicidal thought or drug abuse in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in positive caregiving experience before and after the intervention | T0 (baseline) and (T1) immediately post-intervention
  The Change in caregivers' positive caregiving experience will be measured with the Chinese version of Positive Aspect of Caregiving scale (PAC). The PAC contains 11 items with 5-point Likert scale for all items responses. Scores for each items will be summed to compute a total score which ranges from 11 to 55, with higher scores indicating a more positive self-perceptions of caregiving.
Change in stress before and after the intervention | T0 (baseline) and (T1) immediately post-intervention
  The change in caregivers' stress will be measured with the Chinese version of Perceived Stress Scale (PSS). The PSS contains 10 items with 5-point Likert-type scale rating from 0 (never) to 4 (very often). Scores for each items will be summed up to create a total score. The total score is ranged from 0-40, with higher score representing a higher level of perceived stress.
Change in caregivers' burden before and after the intervention | T0 (baseline) and (T1) immediately post-intervention
  The change of caregiver's burden (only on caregivers) will be measured with the Chinese version of Zarit Burden Interview (ZBI). The scale comprises of 22 items including factors most frequently mentioned by caregivers as problem areas (e.g. caregivers' health, psychological well-being, finances, and social life). Caregivers will be asked to indicate the level of distress caused by each item, ranging from "not at all" to "extremely distressing," on a scale of 0 to 4. A total burden score will be obtained by adding up the scores for each response, with a possible total score ranging from 0 to 88. A higher score indicates greater caregiver distress.
Change in quality of life before and after the intervention | T0 (baseline) and (T1) immediately post-intervention
  The World Health Organization Quality of Life (WHOQOL-OLD) short form will be used to assess the changes of caregivers' quality of life (QOL). The WHOQOL-OLD short form comprises of 6 old aged-specific quality of life items and each item is rated on a 5-point Likert-type scale that ranged from 1 (very dissatisfied) to 5 (very satisfied). Scores for each responses will be summed up to create a total score ranged from 6 to 30. A higher score indicates a better quality of life.
Change in depressive symptoms before and after the intervention | T0 (baseline) and (T1) immediately post-intervention
  Depressive mood changes of caregivers will be measured with the Chinese version of Center for Epidemiological Studies Depression scale (CESD), which is a self-reported measurement on depression containing 20 items. Ratings were based on a 4-point Likert scale ranging from 0 (rarely or none of the time) to 3 (most or all of the time). Items for each responses will be summed up to create a total score ranging from 0 to 60. A higher CESD score indicates a higher level of depression.

SECONDARY OUTCOMES:
Change in cognitive functions of the PWD before and after the interventions | T0 (baseline) and (T1) immediately post-intervention
  Montreal Cognitive Assessment 5-min protocol (MoCA-5-min) will be used to assess changes on PWD' cognitive function over the telephone. The MoCA 5-min protocol consists of four subtests examining five cognitive domains, including attention, verbal learning and memory, executive functions/language, and orientation. Total score of the MoCA 5-min protocol range between 0 and 30, with higher score representing a higher level of cognitive functioning.
Change in behavioral and psychological symptoms of the PWD before and after the intervention | T0 (baseline) and (T1) immediately post-intervention
  Change in behavioural and psychological symptoms of PWD will be measured by the Chinese version of the Neuropsychiatric Inventory-Questionnaire (NPI-Q). NPI-Q is an informant-based instrument that measures the presence and severity of 12 Neuropsychiatric Symptoms (NPS) in patients with dementia and caregivers distress. The caregivers will be asked to identify whether the symptoms of the PWD had been present in the past week, and rate the severity of the symptoms (from a Likert scale ranged from 1 to 3) and the corresponding distress to them (from a Likert scale ranged from 1 to 5). The NPI-Q provides two subscores- total Severity of symptoms and total distress scores. Higher score on these two subscales represent a higher level of symptoms severity of PWD and distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Patrick Kor, Hong Kong, Hong Kong

REFERENCES:
- [Background] Chin WY, Choi EP, Chan KT, Wong CK. The Psychometric Properties of the Center for Epidemiologic Studies Depression Scale in Chinese Primary Care Patients: Factor Structure, Construct Validity, Reliability, Sensitivity and Responsiveness. PLoS One. 2015 Aug 7;10(8):e0135131. doi: 10.1371/journal.pone.0135131. eCollection 2015. PMID 26252739
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] The Practice of Nursing Research: Appraisal, Synthesis, and Generation of Evidence - Seventh edition Grove Susan K The Practice of Nursing Research: Appraisal, Synthesis, and Generation of Evidence - Seventh edition 752pp Elsevier 9781455707362 1455707368 [Formula: see text]. Nurs Stand. 2013 Apr 3;27(31):30. doi: 10.7748/ns2013.04.27.31.30.b1488. PMID 26981669
- [Background] Hamer RM, Simpson PM. Last observation carried forward versus mixed models in the analysis of psychiatric clinical trials. Am J Psychiatry. 2009 Jun;166(6):639-41. doi: 10.1176/appi.ajp.2009.09040458. No abstract available. PMID 19487398
- [Background] Leung DY, Lam TH, Chan SS. Three versions of Perceived Stress Scale: validation in a sample of Chinese cardiac patients who smoke. BMC Public Health. 2010 Aug 25;10:513. doi: 10.1186/1471-2458-10-513. PMID 20735860
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement, 1(3), 385-401. doi:10.1177/014662167700100306
- [Background] Smits CH, de Lange J, Droes RM, Meiland F, Vernooij-Dassen M, Pot AM. Effects of combined intervention programmes for people with dementia living at home and their caregivers: a systematic review. Int J Geriatr Psychiatry. 2007 Dec;22(12):1181-93. doi: 10.1002/gps.1805. PMID 17457793
- [Background] Van't Leven N, Prick AE, Groenewoud JG, Roelofs PD, de Lange J, Pot AM. Dyadic interventions for community-dwelling people with dementia and their family caregivers: a systematic review. Int Psychogeriatr. 2013 Oct;25(10):1581-603. doi: 10.1017/S1041610213000860. Epub 2013 Jul 24. PMID 23883489
- [Background] Wong A, Cheng ST, Lo ES, Kwan PW, Law LS, Chan AY, Wong LK, Mok V. Validity and reliability of the neuropsychiatric inventory questionnaire version in patients with stroke or transient ischemic attack having cognitive impairment. J Geriatr Psychiatry Neurol. 2014 Dec;27(4):247-52. doi: 10.1177/0891988714532017. Epub 2014 Apr 24. PMID 24763069
- [Background] Wong A, Xiong YY, Kwan PW, Chan AY, Lam WW, Wang K, Chu WC, Nyenhuis DL, Nasreddine Z, Wong LK, Mok VC. The validity, reliability and clinical utility of the Hong Kong Montreal Cognitive Assessment (HK-MoCA) in patients with cerebral small vessel disease. Dement Geriatr Cogn Disord. 2009;28(1):81-7. doi: 10.1159/000232589. Epub 2009 Aug 11. PMID 19672065
- [Background] Yu R, Chau PH, McGhee SM, Cheung WL, Chan KC, Cheung SH, Woo J. Trends in prevalence and mortality of dementia in elderly Hong Kong population: projections, disease burden, and implications for long-term care. Int J Alzheimers Dis. 2012;2012:406852. doi: 10.1155/2012/406852. Epub 2012 Oct 14. PMID 23097740
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Chan, T. S., Lam, L. C., & Chiu, H. F. (2005). Validation of the Chinese version of the Zarit Burden Interview. Hong Kong Journal of Psychiatry, 15(1), 9-33.
- [Background] Chau, P. H., McGhee, S. M., Yu, R., Cheung, W. L., Chan, K. C., Cheung, S. H., & Woo, J. (2010). Dementia Trends: Impact of the Ageing Population and Societal Implications for Hong Kong. Hong Kong: The Hong Kong Jockey Club.
- [Derived] Kor PPK, Parial LL, Yu CTK, Liu JYW, Liu DPM, Hon JMK. Effects of a Family Caregiver-Delivered MultiSensory Cognitive Stimulation Intervention for Older People With Dementia During Coronavirus 2019: A Randomized Controlled Trial. Gerontologist. 2024 Feb 1;64(2):gnad054. doi: 10.1093/geront/gnad054. PMID 37179458